CLINICAL TRIAL: NCT01742988
Title: Phase 1 Open Label, Multi-center, Dose-Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of Orally Administered Fimepinostat (CUDC-907), a PI3K and HDAC Inhibitor, in Subjects With Refractory or Relapsed Lymphoma
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetics of Fimepinostat (CUDC-907) in Patients With Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Curis, Inc. (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUDC-907-101
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Lymphoma; Relapsed Lymphoma; Refractory Lymphoma; Relapsed and/or Refractory Lymphoma; Relapsed Ddiffuse Large B-Cell Lymphoma (DLBCL); Refractory Diffuse Large B-Cell Lymphoma (DLBCL); Relapsed and/or Refractory Diffuse Large B-Cell Lymphoma (DLBCL); Double-hit Lymphoma (DHL); Triple-hit Lymphoma (THL); Double-expressor Lymphoma (DEL); High-grade B-cell Lymphoma (HGBL)
Keywords: Lymphoma; DLBCL; MYC; Diffuse Large B-Cell Lymphoma; HGBL; High-grade B-Cell Lymphoma; Double-hit Lymphoma (DHL); Triple-hit Lymphoma (THL); Double-expressor Lymphoma (DEL); P13K; HDAC; Open-Label
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — fimepinostat; CUDC-907; Rituximab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (13):
- Fimepinostat - Continuous Once Daily (Experimental): Fimepinostat 30-60 mg/day
  Interventions: Drug: fimepinostat
- Fimepinostat - 2x/week (Experimental): Fimepinostat 60-240 mg/day
  Interventions: Drug: fimepinostat
- Fimepinostat - 3x/week (Experimental): Fimepinostat 60-180 mg/day
  Interventions: Drug: fimepinostat
- Fimepinostat - 4x/week (Experimental): Fimepinosta 60-180 mg/day
  Interventions: Drug: fimepinostat
- Fimepinostat - 5x/week (Experimental): Fimepinostat 60-180 mg/day
  Interventions: Drug: fimepinostat
- Fimepinostat - Expansion 5x/week (Experimental): Fimepinostat 60 mg on the 5 days on/2 days off
  Interventions: Drug: fimepinostat
- Fimepinostat - Expansion 3x/week (Experimental): Fimepinostat 120 mg 3 days on/4 days off
  Interventions: Drug: fimepinostat
- Fimepinostat 60 mg - Combination w/ rituximab (Experimental): Fimepinostat 60 mg 5 days on.2 days off plus rituximab
  Interventions: Drug: fimepinostat; Drug: Rituximab
- Fimepinostat 120 mg - Combination w/ rituximab (Experimental): Fimepinostat 120 mg 3x/week plus rituximab
  Interventions: Drug: fimepinostat; Drug: Rituximab
- Fimepinostat - Biocomparability Arm (Experimental): Biocomparability Arm
  Interventions: Drug: fimepinostat
- Fimepinostat 30 mg - Combination w/ venetoclax (Experimental): Fimepinostat 30 mg 5 days on/2 days off plus venetoclax. Different combinations of dose levels for venetoclax will be explored
  Interventions: Drug: fimepinostat; Drug: venetoclax
- Fimepinostat 60 mg - Combination w/ venetoclax (Experimental): Fimepinostat 60 mg 5 days on/2 days off plus venetoclax. Different combinations of dose levels for venetoclax will be explored
  Interventions: Drug: fimepinostat; Drug: venetoclax
- Fimepinostat - Combination w/ venetoclax and rituximab (Experimental): Fimepinostat and venetoclax dosed at dose levels determined for that combination. Rituximab dosed at 375 mg/m2 IV on Day 1 of each 21 day cycle
  Interventions: Drug: fimepinostat; Drug: Rituximab

INTERVENTIONS:
Drug: fimepinostat
  Other Names: CUDC-907
Drug: Rituximab
  Arms: Fimepinostat - Combination w/ venetoclax and rituximab; Fimepinostat 120 mg - Combination w/ rituximab; Fimepinostat 60 mg - Combination w/ rituximab
Drug: venetoclax
  Arms: Fimepinostat 30 mg - Combination w/ venetoclax; Fimepinostat 60 mg - Combination w/ venetoclax

SUMMARY:
This is a phase 1, open-label, dose-escalation study of fimepinostat (CUDC-907) in patients with relapsed and/or refractory diffuse large B-cell lymphoma (DLBCL), or high-grade B-cell lymphoma (HGBL) with or without MYC and BCL2 alterations. Fimepinostat (CUDC-907) is a multi-targeted agent designed to inhibit phosphoinositide 3-kinase (PI3K)and histone deacetylase (HDAC). The study is designed to assess the safety, the maximum tolerated dose, the recommended phase 2 dose (RP2D), pharmacokinetics and the anti-cancer activity of oral fimepinostat in combination with 1 or more anti-cancer regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with any of the following: Histopathologically confirmed DLBCL or HGBL (i.e., HGBL with MYC, BCL2, and/or BCL6 rearrangements, HGBL, not otherwise specified [NOS], or DLBCL, NOS) that is refractory to, or has relapsed after, treatment with at least 1 prior regimen. Eligible sub-types include DHL, THL, or DEL, as well as DLBCL or HGBL without MYC and/or BCL2 alterations. Criteria for DHL are concurrent MYC translocation+ and BCL2 translocation+ by fluorescence in situ hybridization (FISH) (same criteria for THL, which also includes BCL6 translocation+ by FISH); criteria for DEL are concurrent overexpression of MYC (≥ 40%) and BCL2 (> 50%) by immunohistochemistry (IHC).
* Measurable disease by CT or PET/CT. MRI acceptable as per protocol.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Recovery to Grade 1 or baseline of any toxicity due to prior systemic treatments (excluding alopecia).
* Absolute neutrophil count ≥ 1,000/µL; platelets ≥ 75,000/µL for patients with no bone marrow involvement by malignancy; platelets ≥ 50,000/µL for patients with bone marrow involvement by malignancy.
* Creatinine ≤ 1.5x upper limit of normal (ULN); total bilirubin ≤ 1.5x ULN; AST/ALT ≤ 2.5x ULN.
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Intention to undergo stem cell transplant (SCT) or treatment with chimeric antigen receptor (CAR) T-cell therapy.
* SCT therapy within 100 days prior to starting study treatment.
* Systemic anti-cancer therapy or investigational agent within 3 weeks of study entry, except for nitrosoureas or mitomycin C (6 weeks).
* Other non-cytotoxic anti-cancer therapy or investigational agent within 5 half-lives or 21 days prior to study treatment, whichever is shorter, as long as any drug related toxicities have resolved to Grade 1 or less. Dexamethasone up to 12 mg/d is allowed as supportive therapy and does not exclude participation.
* Contraindication to venetoclax or rituximab.
* Progressive disease during treatment or within 3 months of stopping prior treatment with a BCL2 inhibitor, histone deacetylase (HDAC) inhibitor, or phosphoinositide-3 kinase (PI3k) inhibitor, or prior discontinuation of any of these therapies due to clinically significant toxicity.
* Graft vs. host disease following prior allogeneic transplant within 3 months prior to study treatment.
* Ongoing treatment with chronic immunosuppressants.
* Active CNS lymphoma.
* Known gastrointestinal condition that would interfere with swallowing or the oral absorption or tolerance of fimepinostat.
* Serious infection requiring systemic antibiotic therapy within 14 days prior to study treatment.
* Uncontrolled or severe cardiovascular disease
* Unstable or clinically significant concurrent medical condition.
* Second primary malignancy within 2 years of study entry other than what is specified in the protocol.
* Known HIV positive, hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection.
* Active CMV infection, presence of CMV antigenemia, or evidence of any invasive CMV end organ disease (e.g., CMV colitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-12; Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of oral fimepinostat (CUDC-907) in combination with venetoclax and rituximab | At the end of cycle 1 or 2 (each cycle is 21 days)
  To be evaluated in patients with relapsed and/or refractory (R/R) diffuse large B-cell lymphoma (DLBCL) or high-grade B-cell lymphoma (HGBL). Within any given study arm, the highest dose level studied at which fewer than 2 out of 6 subjects (< 33%) experience a dose limiting toxicity (DLT).
To assess the safety and tolerability of fimepinostat in combination with anti-cancer regimens by evaluating the number of participants with adverse events assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE, v4.0). | 18 months
  Number of participants with adverse events assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE, v4.0).
To evaluate the efficacy of fimepinostat in combination with anti-cancer regimens by evaluating ORR | 24 months
  ORR assessments as measured using Lugano criteria.
To evaluate the efficacy of fimepinostat in combination with anti-cancer regimens by evaluating DOR | 24 months
  DOR assessments as measured using Lugano criteria.

SECONDARY OUTCOMES:
To assess pharmacokinetics (PK) of fimepinostat when administered in combination with anti-cancer regimens as measured by area under the concentration-time curve (AUC). | Pre-dose to 21 - 28 days post dose
  Pharmacokinetic parameters will include area under the concentration-time curve (AUC).
To assess pharmacokinetics (PK) of fimepinostat when administered in combination with anti-cancer regimens as measured by maximum plasma concentration (Cmax). | Pre-dose to 21 - 28 days post dose
  Pharmacokinetic parameters will include maximum plasma concentration (Cmax).
To assess pharmacokinetics (PK) of fimepinostat when administered in combination with anti-cancer regimens as measured by half-life (T1/2). | Pre-dose to 21 - 28 days post dose
  Pharmacokinetic parameters will include half-life (T1/2).
To assess pharmacokinetics (PK) of fimepinostat when administered in combination with anti-cancer regimens as measured by clearance (Cl). | Pre-dose to 21 - 28 days post dose
  Pharmacokinetic parameters will include clearance (Cl).
To assess pharmacokinetics (PK) of fimepinostat when administered in combination with anti-cancer regimens as measured by volume of distribution (Vd). | Pre-dose to 21 - 28 days post dose
  Pharmacokinetic parameters will include volume of distribution (Vd).
To assess PK of venetoclax when administered in combination with fimepinostat as measured by area under the concentration-time curve (AUC). | Pre-dose to 21 - 28 days post dose
  Pharmacokinetic parameters will include area under the concentration-time curve (AUC).
To assess PK of venetoclax when administered in combination with fimepinostat as measured by maximum plasma concentration (Cmax). | Pre-dose to 21 - 28 days post dose
  Pharmacokinetic parameters will include maximum plasma concentration (Cmax).
To assess PK of venetoclax when administered in combination with fimepinostat as measured by half-life (T1/2). | Pre-dose to 21 - 28 days post dose
  Pharmacokinetic parameters will include half-life (T1/2).
To assess PK of venetoclax when administered in combination with fimepinostat as measured by clearance (Cl). | Pre-dose to 21 - 28 days post dose
  Pharmacokinetic parameters will include clearance (Cl).
To assess PK of venetoclax when administered in combination with fimepinostat as measured by volume of distribution (Vd). | Pre-dose to 21 - 28 days post dose
  Pharmacokinetic parameters will include volume of distribution (Vd).
To evaluate the efficacy of fimepinostat in combination with anti-cancer regimens as measured by OS. | 24 months
  OS measured using RECIL 2017 criteria and revised RECIST 1.1.
To evaluate the efficacy of fimepinostat in combination with anti-cancer regimens as measured by PFS. | 24 months
  PFS measured using RECIL 2017 criteria and revised RECIST 1.1.
To evaluate the efficacy of fimepinostat in combination with anti-cancer regimens as measured by ORR. | 24 months
  ORR measured using RECIL 2017 criteria and revised RECIST 1.1.
To evaluate the efficacy of fimepinostat in combination with anti-cancer regimens as measured by DOR. | 24 months
  DOR measured using RECIL 2017 criteria and revised RECIST 1.1.
To evaluate biomarkers of fimepinostat activity | 24 months
  Exploratory biological markers of fimepinostat activity will be assessed in PBMCs, plasma, and tumor and samples to explore biomarkers that correlate with safety and/or efficacy, such as CREBBP/EP300.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Stephenson Cancer Center, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington

REFERENCES:
- [Derived] Oki Y, Kelly KR, Flinn I, Patel MR, Gharavi R, Ma A, Parker J, Hafeez A, Tuck D, Younes A. CUDC-907 in relapsed/refractory diffuse large B-cell lymphoma, including patients with MYC-alterations: results from an expanded phase I trial. Haematologica. 2017 Nov;102(11):1923-1930. doi: 10.3324/haematol.2017.172882. Epub 2017 Aug 31. PMID 28860342
- [Derived] Younes A, Berdeja JG, Patel MR, Flinn I, Gerecitano JF, Neelapu SS, Kelly KR, Copeland AR, Akins A, Clancy MS, Gong L, Wang J, Ma A, Viner JL, Oki Y. Safety, tolerability, and preliminary activity of CUDC-907, a first-in-class, oral, dual inhibitor of HDAC and PI3K, in patients with relapsed or refractory lymphoma or multiple myeloma: an open-label, dose-escalation, phase 1 trial. Lancet Oncol. 2016 May;17(5):622-31. doi: 10.1016/S1470-2045(15)00584-7. Epub 2016 Mar 31. PMID 27049457